CLINICAL TRIAL: NCT06465836
Title: Beni-Suef University Hospital Simplified Conservative Approach for Managing Placenta Accreta Spectrum: RCT
Brief Title: Simplified Conservative Measures in Managing Morbidly Adherent Placenta in Beni-Suef University
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nesreen Abdel Fattah Abdullah Shehata (Other)
Responsible Party: Sponsor-Investigator, Nesreen Abdel Fattah Abdullah Shehata, Professor, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Morbidly adherent placenta
Record Dates: First submitted 2024-05-12; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups. One of two intraoperative surgical interventions that will be evolved during the study period:
  Group A: In which 86 patients will have bilateral uterine artery ligations as described by the O- lreay technique in addition to standard conservative methods. The stitches were tied securely anteriorly.
  Group B: which will include 86 patients we will do our simplified approach which include;
  * After placental separation; try to grasp lower segment, or cervical flap.
  * Close uterine cavity by continuous vicryl no 1 suture.
  * Do 3 to 4 mattress sutures as the second layer of the uterus.
  * Do uterine ligation with compression of the lower uterine segment (Modification of O, lreay suture).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done by online research randomizer as follows (https://www.randomizer.org/about/ ):
  2 Sets of 86 Unique Numbers Per Set Range: From 1 to 172
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- O- lreay technique group (Other): Group A: In which 86 patients will have bilateral uterine artery ligations as described by O- lreay technique in addition to standard conservative methods. Briefly, two large vicryl stitches were passed using a large-sized needle below and lateral to the lower edge of the uterine incision angle in an anteroposterior direction and then redirected from back to the front through the avascular window in the posterior leaf of the broad ligament just lateral to the uterine border taking care to avoid injury to bowel posteriorly or bladder/ureter anteriorly. The stitches were tied securely anteriorly
  Interventions: Procedure: O, lreay suture
- Modified O- lreay technique group (Other): Group B: which will include 86 patients we will do our simplified approach which includes;
  * After placental separation; try to grasp the lower segment or cervical flap.
  * Close uterine cavity by continuous vicryl no 1 suture.
  * Do 3 to 4 mattress sutures as the second layer of the uterus.
  * Do uterine ligation with compression of the lower uterine segment (Modification of O, lreay suture) as demonstrated below:
    1. Pack Douglas- pouch with a towel.
    2. Straight the used vicryl needle mostly no 1.
    3. Try to compress and approximate anterior and posterior uterine walls.
    4. Start from anterior to posterior 3- 4 cm medial to lateral uterine margin and then pass from posterior to anterior through avascular area in the broad ligament.
  Interventions: Procedure: modified O, lreay suture

INTERVENTIONS:
Procedure: O, lreay suture — bilateral uterine artery ligations as described by O- lreay technique in addition to standard conservative methods. Briefly two large vicryl stitches were passed using a large sized needle below and lateral to the lower edge of the uterine incision angle in anteroposterior direction and then redirected from back to the front through avascular window in the posterior leaf of the broad ligament just lateral to the uterine border taking care to avoid injury to bowel posteriorly or bladder/ureter anteriorly. The stitches were tied securely anteriorly
  Arms: O- lreay technique group
Procedure: modified O, lreay suture — 1. Pack Douglas- pouch with a towel.
  2. Straight the used vicryl needle mostly no 1.
  3. Try to compress and approximate anterior and posterior uterine walls.
  4. Start from anterior to posterior 3- 4 cm medial to lateral uterine margin and then pass from posterior to anterior through avascular area in the broad ligament. And we repeat the procedure on the other side. We can repeat this method of uterine ligation at another different plane if needed.
  Arms: Modified O- lreay technique group

SUMMARY:
To evaluate the efficacy of modified uterine artery ligation and myometrial compression as a conservative measure in improving the prognosis of the morbidly adherent placenta.

DETAILED DESCRIPTION:
According to the International Federation of Gynecology and Obstetrics (FIGO) guidelines, the principal surgical strategy to prevent excessive bleeding related to placenta accreta syndrome is to leave the placenta in situ and perform a primary peripartum hysterectomy at delivery. A hysterectomy may not be preferred by patients wishing to preserve fertility and is detrimental to multiple aspects of the pelvic floor, bowel, and physical functions.

Surgical principles in placenta accreta syndrome include avoiding disruption of the hypervascular placenta, stepwise devascularization, early and comprehensive blood product transfusion, and judicious use of interventional radiologic techniques such as vascular embolization.

Conservative management describes any approach whereby hysterectomy is avoided

ELIGIBILITY:
Inclusion Criteria:

* Gestational age more than 28 weeks as determined by LMP and ultrasound.
* Placenta previa as confirmed by ultrasound.
* Clinically stable with no or mild vaginal bleeding.
* No evidence of fetal compromise.
* Patient consent.

Exclusion Criteria:

* Vaginal bleeding
* Medical disorders

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Amount of blood loss | 6 hours postoperatively
  The primary outcome for the study is the total volume of blood loss in the intra and postoperative period.

SECONDARY OUTCOMES:
Maternal morbidity | 24 hours post operatively
  Coagulopathy, need for massive blood transfusion (> 4 units), length of hospital stay, and visceral injuries ICU admission and post-operative pain.
Maternal mortality | 24 hours postoperatively
  Maternal death

OTHER OUTCOMES:
Gynecological conditions | 6 months
  Gynecological complications as amenorrhea, intrauterine adhesions and niche formation.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Cairo, Egypt